CLINICAL TRIAL: NCT00901953
Title: Do Migrainous Vertigo Patients Have More Hypersensitivity in Their Vestibular System Than Migraine Patients Without Vertigo?
Brief Title: Vestibular System in Migrainous Vertigo Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Bergen (Other)
Collaborators: Sorlandet Hospital HF (Other Government)
Responsible Party: Marion Ingeborg Boldingh, Departement of Neurology, Sørlandet Hospital HF , Kristiansand, Norway
Other Study IDs: 2.2006.3376
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Migraine Disorders; Migraine Variant; Episodic Recurrent Vertigo
Keywords: migraine; migrainous vertigo; vestibular evoked myogenic potentials; vestibular function test; vestibular disorders
MeSH Terms: conditions — Migraine Disorders; Vestibular Neuronitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: migrainous vertigo
- 2: migraine without vertigo

SUMMARY:
Do migrainous vertigo patients have more pathology in their vestibular system than migraine patients without vertigo?

The aim of this study is to compare the vestibular system of migraine patients with and without vertigo in the symptom-free period by vestibular function tests, videonystagmography, vestibular evoked myogenic potentials, and subjective visual vertical.

ELIGIBILITY:
Inclusion Criteria:

* migraine according to IHS criteria
* migrainous vertigo according to the Neuhauser-criteria

Exclusion Criteria:

* no history of other neurological, vestibular, opthalmologic and ENT disorders
* no medications that could possibly influence test results
* intact hearing measured by audiometry
* pregnancy

Ages: 16 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Migraine patients: primary care clinic
  Migrainous vertigo patients: Neurological outpatients clinic, Sorlandet Hospital HF, Kristiansand and Spesialistsenteret, Tollbodgata 4, Kristiansand.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Differences in vestibular function | Symptomfree interval

SECONDARY OUTCOMES:
Differences in hypersensitivity | Symptomfree interval

CONTACTS AND LOCATIONS:
Overall Officials: Åse Mygland, PhD, Principal Investigator — Institute of clinical medicine, university of Bergen, Norway
Locations (1):
- Dept. of neurology, Sørlandet Hospital HF, Kristiansand, Kristiansand, Norway